CLINICAL TRIAL: NCT04446052
Title: Phase III Study Priming With rhu_GM-CSF and of Three Induction Regimens in Adult Patients (55 and Over) With Acute Non-Lymphocytic Leukemia
Brief Title: Phase III rhu_GM-CSF + 3 Induction Regimens in Adults With Acute Non-Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E3993
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Adult Patients (Over 55) With Acute Non-Lymphocytic Leukemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- GM-CSF priming (Active Comparator)
  Interventions: Drug: GM-CSF priming

INTERVENTIONS:
Drug: GM-CSF priming
  Arms: GM-CSF priming
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Phase III Study of Priming with Granulocyte-Macrophage Colony Stimulating Factor (rhu-GM-CSF) and ofThree Induction Regimens in Adult Patients (Over 55) with Acute Non-Lymphocytic Leukemia

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute non-lymphocytic leukemia are eligible for the study.

Exclusion Criteria:

* N/A

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 1993-05-21 (Actual); Primary Completion 2002-07-10 (Actual); Study Completion 2002-07-10 (Actual)

PRIMARY OUTCOMES:
complete remission rates | 3 years